CLINICAL TRIAL: NCT03980132
Title: Randomized Clinical Trial, Blinded for the Researcher and Multicenter, to Evaluate the Efficacy and Safety of Preoperative Preparation With Lugol Solution in Euthyroid Patients With Graves-Basedow Disease.
Brief Title: Preoperative Preparation With Lugol Solution in Patients With Graves-Basedow Disease.
Acronym: LIGRADIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jesús María Villar del Moral (Other)
Responsible Party: Sponsor-Investigator, Jesús María Villar del Moral, Head of General and Digestive Surgery - H. U. Virgen de las Nieves, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIGRADIS
Record Dates: First submitted 2019-05-30; First posted 2019-06-10 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hyperthyroidism, Autoimmune
Keywords: Thyroid Surgery; Grave' Disease; Lugol Solution
MeSH Terms: conditions — Graves Disease | interventions — iodine potassium iodide

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative Lugol Solution preparation (Experimental): Patients will receive Lugol Solution preparation for 10 days before thyroidectomy
  Interventions: Drug: Lugols Strong Iodine
- No preparation (No Intervention): Patients will not receive preparation before thyroidectomy

INTERVENTIONS:
Drug: Lugols Strong Iodine — 5 L.I. drops / 8 hours for 10 days before surgery
  Arms: Preoperative Lugol Solution preparation

SUMMARY:
Currently, both the American Thyroid Association and the European Thyroid Association recommend the use of Lugol Solution (LS) in the preparation of patients undergoing thyroidectomy for Graves' disease (GD), but their recommendations are based on a low level of evidence. This means that its use is not generalized among the different endocrine surgery units.

Methods:

Study population: 270 patients (135 patients in each arms) undergoing total thyroidectomy (TT) due to GD in Spanish hospitals, which perform a minimum of 100 thyroidectomies a year, at least 10 of them for GD.

Variables:

Preoperative variables

* Demographic variables: birthdate, gender and ethnicity.
* Drugs allergies. Allergy to iodine.
* Personal history and usual treatment.
* Aspects related to the GD: date of diagnosis, use of AT drugs and/or radioiodine, existence of ophthalmopathy, existence of cervical compression symptoms and indication of surgery.
* Physical exploration: body mass index, pulse at rest and blood pressure and cervical palpation.
* Laboratory tests: hematocrit, leukocytes, neutrophils, platelets, international normalized ratio(INR), creatinine, potassium, total calcium, albumin, total proteins, parathormone (PTH), 25-hydroxide-vitamin D, free T4 and / or free T3, TSH, thyroid stimulating immunoglobulin (TSI).
* Classification of the anesthetic risk of ASA.
* Cervical ultrasound: existence of thyroid nodules and volume of the thyroid.
* Mobility of the vocal cords evaluated by laryngoscopy.
* Compliance with assigned treatment: the patient assigned to the LS arm must have consumed at least 80% of the total dose indicated.

Intraoperative variables

* Surgical time.
* Antibiotic prophylaxis
* Intraoperative hemorrhage.
* Thyroidectomy Difficulty Scale.
* Loss of electromyographic signal during neural intraoperative monitorization.
* Accidental parathyroidectomy.
* Section or obvious lesion of the recurrent laryngeal nerve.
* Trachea or esophagus perforation.
* Weight of the gland.
* Electrosurgical hemostasis system used during the intervention.
* Maneuvers used to check hemostasis.
* Hemostats used during the intervention.
* Use of drainage.
* Definitive surgical technique: TT, unilateral or bilateral subtotal thyroidectomy or hemithyroidectomy.

Postoperative variables

* Early complications: hypoparathyroidism, paralysis of the recurrent laryngeal nerve, postoperative hematoma, surgical site infection or death.
* Debit for surgical drains.
* Postoperative hospital long of stay.
* Anatomopathological variables: histological diagnosis compatible with GD and existence of parathyroid glands in the surgical specimen.
* Long-term complications: hypocalcemia and/or permanent vocal cord paralysis longer than 6 months

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria will be eligible:

* The age of the patient must be over 18 years of age.
* The patient or his / her tutor, in cases where this is the case, has the capacity to understand the study and agrees to participate in it, by signing the corresponding informed consent document.
* Patients who have been diagnosed with GD, defined as the existence of hyperthyroidism (TSH < lower limit of laboratory normality associated with TSI > upper limit of laboratory normality) that present ultrasonographic data (diffuse vascularization increase) and / or scintigraphy (diffuse uptake of the radioisotope) compatible with GD.
* Euthyroid patients (free T4 and / or free T3 within the normal range of the laboratory) at the time of randomization, and under treatment with AT drugs (propylthiouracil, carbimazole or methimazole).
* The patient must be proposed for total thyroidectomy, using a transcervical approach.

Exclusion Criteria:

The participant can not participate in the study if he / she presents any of the following circumstances:

* Prior cervicotomy by surgical intervention on the thyroid or parathyroid gland.
* Associated hyperparathyroidism that requires associating a parathyroidectomy in the same surgical act.
* Associated thyroid cancer that requires adding a lymph node dissection of the central or lateral compartment in the same surgical time.
* Iodine allergy.
* Consumption of lithium or amiodarone between randomization and administration of LS.
* Patients with category IV of the anesthetic risk classification of the American Society of Anesthesiologists (ASA).
* Women who breastfeed during the administration of the LS or in the month after it.
* Preoperative palsy of a vocal cord verified by laryngoscopy.
* Surgery performed by training specialists, or by staff not specifically dedicated to endocrine surgery.
* Surgery not performed under general anesthesia.
* Endoscopic surgery, video assisted or by remote approach.
* Surgery performed in out-patient settings.
* Current drug consumption or alcohol abuse that could interfere with meeting the study requirements.
* Participation in any other trial with medications in the month prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days after surgery
  To analyze whether, in euthyroid patients undergoing TT due to GD, preoperative non-preparation with LS increases the appearance of postoperative complications compared to the use of LS preparation. The main variable will be the rate of postoperative complication: hypoparathyroidism, recurrent laryngeal nerve injury, hematoma, surgical site infection or death.

SECONDARY OUTCOMES:
Surgical difficulty | Intraoperatively
  Score of the difficulty of the surgery by the surgeon through the Thyroidectomy Difficulty Scale.
Intraoperative hemorrhage | Intraoperatively
  Amount of blood lost during the thyroidectomy in dL.
Surgical time. | Intraoperatively.
  Time from surgical incision to skin closure in minutes.
Intraoperative neuromonitoring. | Intraoperatively.
  Rate of patients with loss of electromyographic signal during intraoperative neuromonitoring.
Postoperative Long of Stay | 30 days after surgery
  Days to hospital discharge after surgery.
Readmissions | 30 days after surgery.
  Rate of readmissions.
Permanent complications | 180 days after surgery
  Rate of patients with permanent complications, including hypoparathyroidism or recurrent laryngeal nerve injury.
Adverse events | 180 days after surgery
  Number of patients with an adverse event after administration of Lugol solution.

CONTACTS AND LOCATIONS:
Locations (21):
- Spain (21):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Donostia, San Sebastián, Guipúzcoa
  - Hospital Clínico Universitario, Santiago de Compostela, La Coruña
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Hospital Universitario del Mar, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de La princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Munoz de Nova JL, Franch-Arcas G, Mejia-Abril GP, Flores-Ruiz ME, Munoz-Perez N, Pintos-Sanchez E, Guadarrama Gonzalez FJ, Valdes de Anca A, Mercader-Cidoncha E, de la Quintana-Basarrate A, Osorio-Silla I, Ros-Lopez S, Gallego-Otaegui L, Santos-Molina E, Martinez-Nieto C, Gamborino-Carames E, Artes-Caselles M, Lorente-Poch L, Garcia-Carrillo M, Moreno-Llorente P, Marin-Velarde C, Ortega-Serrano J, Martos-Martinez JM, Vidal-Perez O, Luengo-Pierrard P, Villar-Del-Moral JM. Efficacy and safety of preoperative preparation with Lugol's iodine solution in euthyroid patients with Graves' disease (LIGRADIS Trial): Study protocol for a multicenter randomized trial. Contemp Clin Trials Commun. 2021 Jun 15;22:100806. doi: 10.1016/j.conctc.2021.100806. eCollection 2021 Jun. PMID 34195471